CLINICAL TRIAL: NCT04167189
Title: Prevalence of Lidocaine Ineffectiveness in Those With Hard-to-treat ADHD
Brief Title: Observational Study to Assess the Frequency of Lidocaine Ineffectiveness in Hard-to-treat ADHD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: PhenoSolve, LLC (Industry)
Collaborators: NeurAbilities (formerly CRCNJ) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-01A
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Using a taste-based test before and after the application of lidocaine gel to the tongue, we will assess the degree to which lidocaine is effective at blocking taste in those with hard-to-treat ADHD
Masking Description: The scoring of the lidocaine test is masked, using the coded identity of the tastes. The tastes will be assessed in random order. The subjects and other study personnel will be told not to discuss what the subject could or couldn't taste. Scoring will not be shared with the testing site until all testing is complete.
  This is one of the last studies with an IRB for each arm and site. Hence it appears to be a single arm, but the other arms are separately registered with ClinicalTrials.gov
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Observational study of prevalence in hard-to-treat ADHD (Other): Subjects will be tested with lidocaine gel.
  Interventions: Drug: Lidocaine gel

INTERVENTIONS:
Drug: Lidocaine gel — Septodont 5% oral lidocaine gel (NDC 0362-0221-10), 75 mg
  Other Names: Intervention

SUMMARY:
This work will assess the prevalence in hard-to-treat ADHD of the ineffectiveness of the anesthetic Lidocaine.

DETAILED DESCRIPTION:
Using a non-invasive, pain-free, taste-based approach to assess lidocaine effectiveness, the study will assess the frequency of ineffectiveness in the target population.

ELIGIBILITY:
Inclusion Criteria: ADHD

Exclusion Criteria for both arms:

1. known adverse reactions to lidocaine
2. epilepsy, IQ <80, severe head trauma, birth weight <2270 grams, and severe autism;
3. treatment currently with potassium or potassium-elevating drugs such as renin-angiotensin-aldosterone blockers;
4. generalized anxiety disorders (but dental-specific anxiety will not be an exclusion because many of these individuals may be ones with anxiety because of painful dental experiences with lidocaine ineffectiveness);
5. mouth sores;
6. Ehlers Danlos syndrome, and
7. red hair.

Ages: 7 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Segal, MD PhD, Principal Investigator — PhenoSolve, LLC
Locations (1):
- NeurAbilitis, Voorhees Township, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to submit for publication descriptions of what was accomplished, and the evaluations as described in the study, including the incidence of lidocaine ineffectiveness in those with ADHD and in the general population.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months

REFERENCES:
- [Background] Infante MA, Moore EM, Nguyen TT, Fourligas N, Mattson SN, Riley EP. Objective assessment of ADHD core symptoms in children with heavy prenatal alcohol exposure. Physiol Behav. 2015 Sep 1;148:45-50. doi: 10.1016/j.physbeh.2014.10.014. Epub 2014 Oct 23. PMID 25447751
- [Background] Levitt JO. Practical aspects in the management of hypokalemic periodic paralysis. J Transl Med. 2008 Apr 21;6:18. doi: 10.1186/1479-5876-6-18. PMID 18426576
- [Background] Nakai Y, Milgrom P, Mancl L, Coldwell SE, Domoto PK, Ramsay DS. Effectiveness of local anesthesia in pediatric dental practice. J Am Dent Assoc. 2000 Dec;131(12):1699-705. doi: 10.14219/jada.archive.2000.0115. PMID 11143733
- [Background] Segal MM. We cannot say whether attention deficit hyperactivity disorder exists, but we can find its molecular mechanisms. Pediatr Neurol. 2014 Jul;51(1):15-6. doi: 10.1016/j.pediatrneurol.2014.04.014. Epub 2014 Apr 18. No abstract available. PMID 24938135
- [Background] Segal MM, Rogers GF, Needleman HL, Chapman CA. Hypokalemic sensory overstimulation. J Child Neurol. 2007 Dec;22(12):1408-10. doi: 10.1177/0883073807307095. PMID 18174562
- [Background] Segal MM, Douglas AF. Late sodium channel openings underlying epileptiform activity are preferentially diminished by the anticonvulsant phenytoin. J Neurophysiol. 1997 Jun;77(6):3021-34. doi: 10.1152/jn.1997.77.6.3021. PMID 9212254
- [Background] Teicher MH, Polcari A, Fourligas N, Vitaliano G, Navalta CP. Hyperactivity persists in male and female adults with ADHD and remains a highly discriminative feature of the disorder: a case-control study. BMC Psychiatry. 2012 Nov 7;12:190. doi: 10.1186/1471-244X-12-190. PMID 23134619
- See also: Saul R (2014) "ADHD Does Not Exist". HarperCollins — https://www.amazon.com/ADHD-Does-Not-Exist-Hyperactivity/dp/006226673X
- See also: Rozanski RJ, Primosch RE, Courts FJ (1988). Clinical efficacy of 1 and 2% solutions of lidocaine. Pediatr Dent.10:287-90 — https://pdfs.semanticscholar.org/1778/f693dc7dd257ab98a96b5bf03408d9cef3eb.pdf
- See also: Segal MM, Jurkat-Rott K, Levitt J, Lehmann-Horn F (2014) Hypokalemic periodic paralysis - an owner's manual — https://www.uni-ulm.de/fileadmin/website_uni_ulm/med.inst.040/Dokumente/owner.html
- See also: Segal MM (2015) Devices, Kits, and Methods for Determining Sensitivity to Anesthetics. US Patent Filing 62/210,747, Filed 09/14/2015 — https://patents.google.com/patent/WO2017035470A1/en
- See also: Companion study — https://clinicaltrials.gov/ct2/show/NCT03563573

RESULTS

PARTICIPANT FLOW:
Groups:
- Hard-to-treat ADHD: Subjects will be tested with Septodont 5% oral lidocaine gel (NDC 0362-0221-10), 75 mg pre-measured by compounding pharmacy and dispensed into blister pack
Period: Overall Study
Arm/Group | Hard-to-treat ADHD
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study
Arm/Group | Hard-to-treat ADHD
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
Hard-to-treat ADHD (does not respond to available ADHD drugs) [Count of Participants; unit: Participants] | 28

OUTCOME MEASURES:

1. Primary Outcome: Observational Study: Number of Participants With Lidocaine Ineffectiveness by Taste Test in Hard-to-treat ADHD
Description: Subjects will be asked to identify each taste and its intensity.
Time Frame: on day of testing, approximately 30 minutes for clinic visit
Population: Study population vs. previously published studies in pediatric populations (Nakai et al, 2000)
Measure: Count of Participants; unit: Participants
Arm/Group | Hard-to-treat ADHD
Number analyzed (Participants) | 28
Participants
  Lidocaine effective (got numb) | 1
  Lidocaine ineffective (did not get numb) | 27

ADVERSE EVENTS:
Time Frame: on day of testing, approximately 60 minutes for clinic visit
Arm/Group | Hard-to-treat ADHD
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
This was an observational study without controls, as there were no controls available at the site. NeurAbilities is a clinic dedicated to treating patients with neurological diagnoses. To do statistics, the study will need to be repeated at a site that can provide controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT04167189/Prot_000.pdf